CLINICAL TRIAL: NCT01221324
Title: Diagnostic Value of C-reactive Protein and White Blood Cell Counts for Early Detection of Inflammatory Complications After Open Resection of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Ignazio Tarantino, M.D., Cantonal Hospital of St. Gallen
Other Study IDs: EKSG10/126
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Given Indication for Open Resection of Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients after open resection of colorectal cancer

SUMMARY:
Although widely used, there is a lack of evidence concerning diagnostic value of C-reactive protein (CRP) and white blood cell counts (WBC) in the postoperative course. The aim of this study was to evaluate the diagnostic accuracy of CRP and WBC for postoperative inflammatory complications after open resection of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* all patients with resection of colorectal cancer

Exclusion Criteria:

* lack of measurement of C-reactive protein
* lack of measurement of white blood cell counts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given indication for resection of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
postoperative inflammatory complications | 30 days

SECONDARY OUTCOMES:
Anastomotic leakage | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Rene Warschkow, MD, Principal Investigator — Cantonal Hospital of St. Gallen

REFERENCES:
- [Background] Warschkow R, Tarantino I, Torzewski M, Naf F, Lange J, Steffen T. Diagnostic accuracy of C-reactive protein and white blood cell counts in the early detection of inflammatory complications after open resection of colorectal cancer: a retrospective study of 1,187 patients. Int J Colorectal Dis. 2011 Nov;26(11):1405-13. doi: 10.1007/s00384-011-1262-0. Epub 2011 Jun 24. PMID 21701807